CLINICAL TRIAL: NCT03354494
Title: Desogestrel (DSG) and Corifolitropin (FSH-CTP) Alfa for Ovarian Stimulation in Donors
Status: Completed | Type: Observational
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Dr. Francisca Martínez, MD PhD, Fundacion Dexeus
Other Study IDs: SMD-DSG-2017-15
Record Dates: First submitted 2017-09-28; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Controlled Ovaria Stimulation
Keywords: Oocyte donors; Ovarian stimulation; Desogestrel; Corifolitropina alfa; Gonadotropins
MeSH Terms: interventions — Desogestrel; follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DSG-CTP
  Interventions: Drug: Desogestrel (DSG) and Corifolitropin (FSH-CTP) Alfa

INTERVENTIONS:
Drug: Desogestrel (DSG) and Corifolitropin (FSH-CTP) Alfa

SUMMARY:
Currently, controlled ovarian stimulation (COS) in oocyte donors is performed by daily injections of gonadotropins( recombinant FSH) plus a GnRH Antagonist usually form 5th-6th stimulation day until ovulation induction with a bolus of another injection of a gonadotropin-releasing hormone (GnRH) Agonist. Injections of the GnRH Antagonist avoid untimely luteinizing hormone (LH) surge and spontaneous ovulation prior to follicular aspiration. There is a preparation of long-acting recombinant follicle stimulating hormone (rFSH= (corifollitropin alfa (FSH-CTP), Elonva®, MSD), that allows that a single subcutaneous injection substitutes the first 7 days of daily gonadotropin injections. On the other hand, a contraceptive oral progesterone only( Desogestrel, DSG) is available for contraception, avoiding the LH surge.

In donors, by administering a single injection of FSH-CTP and oral desogestrel since the first menstruation day, the total number of injections administered is reduced and less discomfort is experienced without adverse impact on ovarian response.

Other authors have reported good results using similar synthetic progestins (Medroxyprogesterone, dihydrogesterone, and natural progesterone).

No description of the hormonal and ovarian response under this protocol has been published. Direct comparison between this novel protocol and the classical GnRH- antagonist plus daily gonadotropins has not been reported.

ELIGIBILITY:
Inclusion Criteria:

-Fulfilling inclusión medical and legal criteria (RD - Spanish law adapting european rule-9/2014)

* Who had had undergone previously convencional COS (controlled ovarian stimulation) with FSH-CTP and daily antagonist injections
* Given signed consent form.

Exclusion Criteria:

* Previous low response to COS
* Previous ovarian hyperstimulation syndrome.
* Ovarian cysts.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: - Population: donors (18-35 ) from candidates of Donor program
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Total dose of gonadotrophins | At the end of stimulation treatment period (from day of corifollitropin administration until the day of triggering) ) an average 10 days after beginning treatment
  Sum of gonadotrophins dose
Oocyte retrieved | Oocyte retrieval day an average 10 days after beginning treatment
  Number of oocyte retrieved

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez F, Boada M, Coroleu B, Clua E, Parera N, Rodriguez I, Barri PN. A prospective trial comparing oocyte donor ovarian response and recipient pregnancy rates between suppression with gonadotrophin-releasing hormone agonist (GnRHa) alone and dual suppression with a contraceptive vaginal ring and GnRH. Hum Reprod. 2006 Aug;21(8):2121-5. doi: 10.1093/humrep/del121. Epub 2006 Apr 21. PMID 16632462
- [Background] Martinez F, Clua E, Santmarti P, Boada M, Rodriguez I, Coroleu B. Randomized, comparative pilot study of pituitary suppression with depot leuprorelin versus cetrorelix acetate 3 mg in gonadotropin stimulation protocols for oocyte donors. Fertil Steril. 2010 Nov;94(6):2433-6. doi: 10.1016/j.fertnstert.2010.02.059. Epub 2010 Apr 28. PMID 20430379
- [Background] Requena A, Cruz M, Collado D, Izquierdo A, Ballesteros A, Munoz M, Garcia-Velasco JA. Evaluation of the degree of satisfaction in oocyte donors using sustained-release FSH corifollitropin alpha. Reprod Biomed Online. 2013 Mar;26(3):253-9. doi: 10.1016/j.rbmo.2012.11.015. Epub 2012 Dec 5. PMID 23352098
- See also: Related Info — http://www.dexeus.com